CLINICAL TRIAL: NCT03646929
Title: Motor Evoked Potentials With Modified Facilitation Technique: Normative Data and Reliability in Healthy Individuals and Comparison of Sensitivity and Specificity With Standard Technique in Patients With Multiple Sclerosis
Brief Title: Motor Evoked Potentials With Modified Facilitation Technique
Acronym: EP-F
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 2017-01893; me18Hardmeier
Record Dates: First submitted 2018-08-22; First posted 2018-08-24 (Actual); Last update posted 2021-05-05 (Actual); Status verified 2021-05

CONDITIONS: Multiple Sclerosis
Keywords: facilitation technique; multimodal evoked potentials (mmEP) in multiple sclerosis; motor evoked potential (MEP) in multiple sclerosis
MeSH Terms: conditions — Multiple Sclerosis; Microcephaly, microphthalmia, ectrodactyly of lower limbs, and prognathism

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- healthy individuals and patients with multiple sclerosis (Other): MEP in healthy individuals and patients with multiple sclerosis are measured using standard facilitation technique
  Interventions: Diagnostic Test: MEP using standard facilitation technique
- patients with multiple sclerosis (Other): MEP in patients with multiple sclerosis are measured using modified facilitation technique
  Interventions: Diagnostic Test: MEP using standard facilitation technique; Diagnostic Test: MEP using modified facilitation technique

INTERVENTIONS:
Diagnostic Test: MEP using standard facilitation technique — measuring of MEP using standard facilitation technique according to the Guidelines of International Federation of Clinical Neurophysiology
Diagnostic Test: MEP using modified facilitation technique — measuring of MEP using modified facilitation technique (application of additional 8-12x magnetic stimuli for arms and legs)
  Arms: patients with multiple sclerosis

SUMMARY:
Investigating the change in Test- Retest- reliability in healthy individuals when applying a modified easy to use facilitation technique compared to standard facilitation technique and analyzing sensitivity and specificity in patients with multiple sclerosis regarding detection of pathologic results

ELIGIBILITY:
Inclusion Criteria for healthy individuals:

* Ability to understand the purpose and risks of the study, provide signed and dated informed consent
* Between 18 and 65 year of age
* No neurologic or psychiatric comorbidity requiring continous treatment
* No previous damage of central nervous System

Inclusion Criteria for patients:

* Ability to understand the purpose and risks of the study, provide signed and dated informed consent
* Between 18 and 65 year of age
* patients with inflammatory diseases of the central nervous system (CNS) or multiple sclerosis appointed for routine MEP diagnostic at the Department of Clinical Neurophysiology, University Hospital Basel

Exclusion Criteria:

* Contraindication for measuring of motoric evoked potentials (MEP): metal implants (pacemaker, stents); known epilepsy oder previous epileptic fit
* Known disease of the peripheral nervous system (polyneuropathy)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 81 (Actual)
Dates: Start 2017-12-20 (Actual); Primary Completion 2019-01-15 (Actual); Study Completion 2019-01-15 (Actual)

PRIMARY OUTCOMES:
Change in Test- Re-Test reliability when using modified facilitation technique (compared to standard facilitation technique) in healthy individuals | measuring time 2 (75 minutes) maximal 1 month later than measuring time 1 (75 minutes)
  Determination of mean intra-individual difference between measuring time 1 and measuring time 2 and calculation of standard deviation
comparison of sensitivity and specificity of modified facilitation technique and standard facilitation technique in patients with multiple sclerosis | 1 measuring time (90 minutes)
  Determination on the basis of the standard values (established in healthy individuals) in how many patients a pathological result with the modified facilitation technique and the standard facilitation technique is present. Using a a cross-tabulation, the sensitivity and specificity of the modified facilitating technique compared to the standard facilitation technique is measured

CONTACTS AND LOCATIONS:
Overall Officials: Martin Hardmeier, PD Dr. med, Principal Investigator — University Hospital, Basel, Switzerland
Locations (1):
- Dep. of Neurology and Clinical Neurophysiology , Hospital of the University of Basel, Basel, Switzerland